CLINICAL TRIAL: NCT04957823
Title: Serum Irisin Level & FDNC5 Genetic Polymorphism Can Predict the Presence &Severity of Coronary Artery Disease in Patients With Type II DM?
Brief Title: Irisin Expression and Gene Polymorphism in Type II Diabetic Patients With and Without CAD
Acronym: CAD
Status: Completed | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Amera Morad Foad, clinical professor, Sohag University
Other Study IDs: Soh-Med-21-06-20
Record Dates: First submitted 2021-07-03; First posted 2021-07-12 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Irisin Gene Polymorphism in Type II Diabetic Patients

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Diseased: type II diabetic patients with documented coronary artery disease.
- Control: type II diabetic patients without coronary artery disease.

SUMMARY:
This is an observertional study aimed at Study the association between the level of irisin expression and (Fibronectin Type III Domain Containing 5 (FDNC5) gene polymorphism and the presence and severity of coronary artery disease in patients with Type II DM.

ELIGIBILITY:
Inclusion Criteria:

* This study will include type II diabetic patients aged between 18 and 45 years old

Exclusion Criteria:

1. Recent acute myocardial infarction.
2. patients with Heart Failure
3. Active infection
4. End stage renal failure (GFR < 30 ml/min) or on dialysis
5. Liver cell failure
6. Athletes or having heavy muscular exercise in the previous 3 days

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: type II diabetic patients with and without coronary artery disease in our center in sohag university hospital.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-04-20 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
Irisin level | 6 months
  detect the serum level of irisin hormone by ELIZA in nanogram/decilitre(ng/dl)
FNDC5 Genotyping | 6 months
  whether homogenetic or heterogenetic

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag uniersity hosoital, Sohag, Egypt

REFERENCES:
- [Derived] Foad AM, Hafez A, Youssef W, Ahmed AE, Altaher AM. Irisin expression and FNDC5 (rs3480) gene polymorphism in type 2 diabetic patients with and without CAD. Arch Physiol Biochem. 2024 Oct;130(5):523-528. doi: 10.1080/13813455.2023.2173785. Epub 2023 Feb 2. PMID 36732920